CLINICAL TRIAL: NCT06107205
Title: A Phase 1, Randomized, Open-Label, Three-Treatment, Three-Period Crossover Study to Assess Bioequivalence and Safety of TTYP01 Tablets to Radicava® Injection, and Radicava ORS® in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence of TTYP01 Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Auzone Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TTYP01-02-2022
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TTYP01 (Active Comparator): Healthy subjects were administered 1 single oral dose of 90 mg TTYP01 (3 tablets of the test drugs, test formulation T)
  Interventions: Drug: TTYP01
- Radicava (Active Comparator): Healthy subjects were administered 1 injection of 60 mg Radicava (reference drug R1, intravenous infusion of 60 mg administered over 60 minutes)
  Interventions: Drug: Radicava
- Radicava ORS (Active Comparator): Healthy subjects were administered 1 single oral dose of 105 mg/5 mL Radicava ORS (reference drug R2)
  Interventions: Drug: Radicava ORS

INTERVENTIONS:
Drug: TTYP01 — 1 single oral dose of 90 mg TTYP01 (3 tablets of the test drugs, test formulation T)
  Other Names: Edaravone tablets
  Arms: TTYP01
Drug: Radicava — 1 injection of 60 mg Radicava (reference drug R1, intravenous infusion of 60 mg administered over 60 minutes)
  Other Names: Edaravone injection
  Arms: Radicava
Drug: Radicava ORS — 1 single oral dose of 105 mg/5 mL Radicava ORS (reference drug R2)
  Other Names: Edaravone ORS
  Arms: Radicava ORS

SUMMARY:
This is a Phase 1, Randomized, Open-Label, Three-Treatment, Three-Period Crossover Study to Assess Bioequivalence and Safety of TTYP01 Tablets to Radicava® Injection, and Radicava ORS® in Healthy Adult Subjects Under Fasting Conditions.The objective is To characterize the bioequivalence、safety and tolerability of TTYP01 tablets and Radicava® injection or Radicava ORS®in healthy adult subjects under fasted conditions.In this study, 30 healthy adult subjects will receive TTYP01, or Radicava, orRadicava ORS in each period according to the randomization sequence.

DETAILED DESCRIPTION:
This is a Phase 1, Randomized, Open-Label, Three-Treatment, Three-Period Crossover Study to Assess Bioequivalence and Safety of TTYP01 Tablets to Radicava® Injection, and Radicava ORS® in Healthy Adult Subjects Under Fasting Conditions.

The Primary objective is To characterize the bioequivalence of TTYP01 tablets (Test) and Radicava® injection (Reference 1) or Radicava ORS® (Reference 2) in healthy adult subjects under fasted conditions.

The secondary objective is To determine the safety and tolerability of TTYP01 tablets (Test), Radicava Injection (Reference 1), and Radicava ORS (Reference 2) in healthy adult subjects under fasted conditions.

In this open-label, randomized, 3-formulation, 3-period, crossover study, 30 healthy adult subjects will receive 1 single oral dose of 90 mg TTYP01 (3 tablets of the test drugs, test formulation T), or 1 injection of 60 mg Radicava (reference drug R1, intravenous infusion of 60 mg administered over 60 minutes), or 1 single oral dose of 105 mg/5 mL Radicava ORS (reference drug R2) after an overnight fast in each period according to the randomization sequence. Subjects will be randomized to 1 of 6 parallel sequences (5 subjects per sequence), with a washout period of at least 96 hours between the periods.

The approximate study period is 6 weeks, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all inclusion criteria at screening (or as noted) to be eligible for study participation, as follows:

1. Informed consent signed and dated by the subject
2. Healthy male and female subjects of any ethnic and racial origin, aged 20 to 45 years, inclusive
3. Female subjects who:

   * Are postmenopausal (defined as a minimum of 12 consecutive months of spontaneous amenorrhea confirmed by a serum follicle-stimulating hormone level > 40 IU/L), or
   * Are surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation), confirmed by medical documentations, or
   * Are of child-bearing potential must agree to use at least 1 highly effective method of contraception from at least 1 month prior to the initiation of the study through 3 months after the final dose, where highly effective methods of contraception include:
   * Intrauterine device
   * Intrauterine system
   * Contraceptive implant
   * Combined injectable contraceptives
   * Hormonal oral contraceptives when used in combination with male condoms with spermicide
   * If a female subject confirms that her male partner(s) has been verified to be clinically sterile (ie, documented infertility or surgical sterilization), this method is acceptable as the only means of contraception

   Note: The following are not acceptable methods of contraception:
   * Periodic sexual abstinence (eg, calendar, ovulation, symptothermal, and post-ovulation methods), declaration of sexual abstinence for the duration of the study, withdrawal, and lactational amenorrhea method
   * Spermicides alone
   * Hormonal oral contraceptives alone
   * Male condoms used in combination with female condoms or
   * Agrees to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.
4. Male subjects who are sexually active and whose partners are females of child-bearing potential, even if surgically sterilized (ie, status post vasectomy), who:

   * Avoid sperm donation during the entire study period and through 90 days after the last dose of study drugs, and
   * Agree to practice effective barrier contraception, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject
5. Body mass index (BMI) of 19 to 30 kg/m2 (inclusive) (BMI = weight (kg)/(height [m])2)
6. Non-smokers (defined as having abstained from tobacco- or nicotine-containing products [eg, cigarettes, chewing tobacco, snuff, nicotine patches, and electronic cigarettes] in the 6 months prior to screening), stable light smokers, and ex-smokers will be included. Stable light and ex-smokers are defined as follows: "A light smoker is defined as someone smoking ≤5 cigarettes per day; an ex-smoker is someone who has completely stopped smoking for at least 3 months."
7. In good health, as determined by the investigator at screening and confirmed at check-in, with no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations
8. Subjects must be willing to understand and able to comply with all research procedures and restrictions, and are able to communicate effectively with researchers.

Exclusion Criteria:

Subjects will not be eligible for study participation if they meet any of the exclusion criteria at screening (or as noted), or will be discontinued at the discretion of the investigator in consultation with the medical monitor if they develop any of the exclusion criteria during the study.

1. History of any hypersensitivity or allergic reaction to active ingredients or excipients of the study drugs (eg, known allergy to bisulfite containing foods such as bottled lemon juice, grape juice, canned fruits, wine, jam, jelly, etc.)
2. Positive test result for infectious diseases at screening or baseline, including human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C virus antibody, and syphilis antibody
3. Positive alcohol test at screening or baseline, or has a history of alcohol abuse (alcohol consumption in excess of 1 standard drink per day for women and 2 standard drinks per day for men; whereby 1 standard drink is equivalent to 12 oz beer [5% alcohol], 5 ounces of wine [12% alcohol], and 1.5 ounces of 80 proof [40% alcohol])
4. Females who are pregnant, planning to become pregnant, or breastfeeding during the study or within 3 months after the study; or have a positive pregnancy test result at screening or check-in
5. Any abnormal physical examination, vital sign, ECG, or laboratory values at screening or check-in that are considered clinically significant by the investigator
6. Special dietary requirements or restrictions and cannot follow a uniform diet
7. History of febrile illness or evidence of active infection within 14 days prior to the first dose
8. Any subject with SARS-CoV-2 infection, based on a rapid test or positive polymerase chain reaction for SARS-CoV-2, or subjects who received the SARS-CoV-2 vaccine within 1 month prior to the first dosing, or plans to have the vaccine within 1 month after the last dose
9. Positive drug screen at screening or check-in, or has a history of drug abuse within the past 5 years
10. Clinically significant interventional therapies (surgery, paracentesis, etc.) within 3 months prior to the study, or plan to have any surgeries during the study
11. Blood loss of non-physiological reasons ≥ 400 mL (ie, trauma, blood collection, blood donation) within 3 months prior to the first dose of study drugs, or plan to donate blood during this study and within 1 month after the last dosing
12. Currently uses more than 5 tobacco products (refer to inclusion criterion 6) per day
13. Received an experimental agent (eg, vaccine, drug, biologic, device, blood product, or medication) within 3 months prior to the first dose of study drugs, or plans to receive another experimental agent during the duration of this study
14. Is unwilling to abstain from alcohol-containing products and xanthine/caffeine-containing products, including any foods and beverages, within 48 hours prior to the first dose
15. Used any over-the-counter medications or prescription drugs (other than hormone replacement therapy, oral contraceptives, or 650 mg acetaminophen/day), nutritional supplements, or herbal medicines within 1 month from screening, unless, in the opinion of the investigator and sponsor, the drug will not interfere with study assessments
16. Abnormal renal function estimated glomerular filtration rate calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation < 90 mL/min/1.73 m2
17. Abnormal QT prolongation of QTcF ≥ 450 msec for males or QTcF ≥ 470 msec for females (confirmed by repeated examination)
18. History of hypokalemia or family history of long QT syndrome
19. Any current or historical conditions that may interfere with the absorption/distribution/metabolism/excretion of the study drugs, in the opinion of the investigator (eg, dysphagia, gastrointestinal diseases)
20. Any clinically relevant acute or chronic medical conditions or diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immune, or dermatologic systems that would pose a risk to subject's safety or interfere with the study assessments, as determined by the investigator
21. Poor venous access (eg, history of difficult blood draws) for blood sample collection or intravenous dosing
22. Any other conditions that would, in the opinion of the investigator, put the subjects at increased risk for participation in this study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
PK Parameters-Area under the plasma concentration-time curve (AUC0-inf) from time 0 extrapolated to infinity of unchanged edaravone after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters- AUC from time 0 to the last measurable non-zero concentration（AUC0-t）of unchanged edaravone after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Maximum observed concentration （Cmax） of unchanged edaravone after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose

SECONDARY OUTCOMES:
PK Parameters-Area under the plasma concentration-time curve (AUC0-inf) from time 0 extrapolated to infinity of sulfate and glucuronide metabolites after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters- AUC from time 0 to the last measurable non-zero concentration（AUC0-t）of sulfate and glucuronide metabolites after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Maximum observed concentration （Cmax） of sulfate and glucuronide metabolites after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters- Time to reach Cmax （Tmax）of unchanged edaravone, sulfate, and glucuronide metabolites after TTYP01, Radicava, and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Apparent terminal elimination half-life （T1/2el）of unchanged edaravone, sulfate, and glucuronide metabolites after TTYP01, Radicava, and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Apparent terminal elimination rate constant （Kel）of unchanged edaravone, sulfate and glucuronide metabolites after TTYP01, Radicava and Radicava ORS administration | up to 48 hours each postdose
PK Parameters -Apparent oral drug clearance (parent drug only) （CL/F）of unchanged edaravone after TTYP01and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Total clearance (CL) of unchanged edaravone after Radicava administration | up to 48 hours each postdose
PK Parameters - Mean residence time (MRT）of unchanged edaravone after Radicava administration | up to 48 hours each postdose
PK Parameters -Apparent volume of distribution Vz/F） of unchanged edaravone after TTYP01and Radicava ORS administration | up to 48 hours each postdose
PK Parameters - Volume of distribution during terminal phase (Vz) of unchanged edaravone after Radicava administration | up to 48 hours each postdose
Incidence and Number of Participants with Adverse events and adverse drug reactions | until the last follow-up visit, up to 6 weeks(including screening and follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Robert. Bass, MD, Principal Investigator — ICON plc
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States